CLINICAL TRIAL: NCT04492111
Title: Bone Remodelling Around Implants With Different Macro-design Placed in Post Extraction Sockets: A CBCT Randomized Controlled Clinical Trial.
Brief Title: X-space Implants in Post-extraction Sites.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Felice Roberto Grassi, Professor, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UniBari
Record Dates: First submitted 2020-07-17; First posted 2020-07-30 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Missing Tooth; Osseointegration Failure of Dental Implant
Keywords: primary stability; dental implant; post-extraction dental implant; dental implant macrodesign; implant failure
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial of parallel design with a 1:1 allocation ratio
Who Masked: Participant, Investigator
Masking Description: Patient not aware of the type of implant. Investigator of clinical conditions not aware of the type of implant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- X-space group (Experimental): Each patient of the experimental group will receive one X-space implant.
  Interventions: Procedure: post-extraction dental implant
- 2P group (Active Comparator): Each patient of the control group will receive one 2P implant. Bone System Cylindric implants. Surface Ecotek.
  Interventions: Procedure: post-extraction dental implant

INTERVENTIONS:
Procedure: post-extraction dental implant — Insertion of a dental implant immediately after tooth extraction.

SUMMARY:
Several recent systematic reviews have highlighted how the macrodesign of dental implants can influence stress distribution and biomechanical and biological behavior in implants immediately inserted in post-extraction sites. Finite element analyzes have confirmed the benefit of the inclination of the implant threads in reducing implant displacement in post-extraction sites, increasing primary stability, and decreasing stress in contact with the trabecular bone.

Other comparative studies have shown that the design of the threads of the implant does not affect the distribution of stress in the surrounding bone.

In view of the need to evaluate the influence of implant macrodesign in the case of implants inserted in post-extraction alveoli, this study will examine the clinical results of two different types of implants with different macrodesigns, with the aim of providing scientific evidence in this regard.

The present study will investigate through a randomized controlled trial the effect of thread macrodesign of X-space implants on primary stability and osseointegration when inserted in post-extraction sites, as compared to cylindric 2P implants.

DETAILED DESCRIPTION:
Objectives Evaluate the clinical and radiological performance of a new implant geometry (X-space) with a central and apical thread designed to increase the contact surface with the alveolar bone and allow a greater insertion torque and better primary stability in post-extraction implants.

The evaluation will be done through:

* Estimation of the difference in terms of dimensional changes of the alveolar bone between the following implants placed in fresh post-extraction sites: (1) X-space (test group), (2) Bone System 2P (control group)
* Estimation of primary stability
* Estimation of implant failure
* Estimation of influences of different clinical factors implant and patient-related to the values of the outcomes.

Expected results The null hypothesis is that the X-space implant is better than the 2P implant. Even in the event of non-statistical significance, factors concerning clinical significance and secondary variables will be assessed in order to determine the efficiency of each of the treatments.

MATERIALS AND METHODS Study design The study will be a randomized clinical trial with two arms, each arm belonging to one of the two intervention groups. The randomization sequence will be computer-generated by an independent statistical specialist.

All the interventions will be performed at the same center by 3 different clinicans following the same protocol. Surgeons will be aware of the type of intervention to be performed only after tooth extraction, therefore immediately before performing the intervention of interest.

The type of intervention will be assigned by means of sealed opaque envelopes that will be open immediately before the intervention.

Patients will be provided with adequate and exhaustive information for participation in the study and each patient must sign a detailed informed consent.

All the interventions performed and the procedures followed in this study are in accordance with the ethical standards of the committee responsible for human experimentation (institutional and national) and with the Helsinki Declaration of 1975, revised in 2000.

Sample size The sample size was determined for a first type error (alpha) 0.05 and a study power of 0.9 (beta 0.1). The reference variable is the dimensional change of the thickness of the vestibular crest (measured at the implant platform level).

The minimal effect of interest assessed from previous studies and the researchers' clinical evaluation was established at 1 mm, while the standard deviation was 0.6 mm.

Considering a 20% loss at follow-up, the sample size required for each group was determined at 15 participants, or 30 participants in all.

References:

1. Wittes J. Sample size calculation for randomized controlled trials. Epidemiol Rev. Vol 24, No. 1, 2002.

Procedures foreseen by the study Thirty implants (15 X-Space and 15 Bone System Cylindrical "2P") of variable diameter and of adequate length will be immediately inserted in the post-extraction sites of thirty patients with therapeutic indications for implantation. The implants (Bone System, Milan) are produced on machining centers and subjected to rigorous cleaning treatments and high precision dimensional checks.

The Ecotek surface of the Bone System implants boasts a long experience of 25 years of clinical applications, Implant surface treatment is obtained by sandblasting with ruby corundum and subsequent etching treatment with acids.

• Surgical protocol In all cases, the extractions will be carried out without lifting the flap and preserving the vestibular wall of the alveolus.

All implants will be inserted at the crest level and will be closed by a screw. The surgical procedure requires insertion into the implant tunnel by means of a controlled torque micromotor (max 50 Ncm), at a speed of 20/25 rpm; for this purpose it is necessary to have a special driver (40120701) inserted in the contra-angle handpiece; for manual insertion with controlled torque, a dynamometric ratchet (CRD) with the relative short (40052401) and standard (40052501) drivers are available.

However, the possibility of insertion with a manual screwdriver is maintained, with the usual tools already used for the other Bone System implants.

The post-extraction site will be closed with a collagen membrane and cross suture.

Data collection methods Variables to be measured (outcomes) Patients will undergo a CT Cone Beam examination immediately after implant insertion and 6 months later to evaluate the morphological and dimensional changes of the alveolar bone horizontally and vertically around the tooth / implant. All the measurements will be carried out in a computerized program which will allow to standardize the repeated measurements.

The measurements on the CT Cone Beam exams and the measurements of the secondary variables will be carried out by an operator not aware of the group to which the patients belong (blind examiner).

Criteria for stopping the study

* Observation of high difference between the techniques, indicating one technique as more efficient than the others or a technique as much less efficient than the other (ethical reason).
* High number of patients lost at follow-up (greater than expected when calculating the sample size).

Criteria for the exit of the subject from the study

* Missing presence at the control at 1 and 3 months (for general evaluation and oral hygiene control)
* Missed presence at check and measures at 6 months
* Lack of collaboration at the oral hygiene level (oral hygiene assessment indices)
* Ongoing presence of periodontal diseases or oral mucous membranes. Ongoing presence of systemic diseases (or related medical therapies) that may influence bone metabolism and tissue healing (e.g. Osteoporosis, corticosteroid therapy, immunodepressive therapies, chemotherapy, radiotherapy, etc.).

Expected duration The foreseeable duration of this study is 18-24 months.

Statistical data analysis The statistical analyzes will be carried out by a statistical analysis expert, on coded and non-identifiable groups. The statistical unit will be the patient.

Descriptive analyzes will be conducted for all demographic variables at the beginning and end of therapy. Mann-Whitney test will be used for statistical comparison analyzes of continuous variables between independent groups. In addition, several multilevel regression analyzes will be conducted to assess the dependence of bone changes on the initial thickness of the vestibular wall and on various patient-related variables. For statistical tests the p-value will be established at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Absence of systemic or local diseases that could compromise implant or prosthetic therapy
* Good periodontal health, assessed by periodontal indices
* Presence of premolar / canine / incisor teeth and with extraction indications and with the presence of two adjacent natural teeth.
* Absence of probing greater than 4mm in the vestibular wall of the crestal bone

Exclusion Criteria:

* CT scan performed in the last 5 years
* Active periodontal diseases
* Heavy smokers (more than 20 cigarettes per day)
* Consumers of high alcohol levels
* Therapy with corticosteroids, immunosuppressive therapies, chemotherapy, radiotherapy, pregnancy
* Lack of collaboration for continuous post-intervention re-evaluations

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Buccal bone dimensional changes | 6 months
  Measurements of buccal bone dimensional changes assessed through a series of linear measurements on two cone-beam (immediately after implant insertion and after 6 months). Measurements will be calibrated using the implant as a reference and will be performed at the marginal bone level, at the central spire level and at the apex level. Outcome will be expressed in mm.
Implant failure | 6 months
  Dental implant loss after insertion. Outcome will be assessed during follow-up checks and confirmed through clinical signs of loss (implant mobility) and intraoral radiograph.

SECONDARY OUTCOMES:
Primary stability | immediately after implant insertion
  Measurement of primary stability immediately after implant insertion through Osttell Mentor and expressed as implant stability quotient (ISQ)

OTHER OUTCOMES:
Complications | During the entire follow-up period- up to 6 months.
  Complications during and after implant insertion assessed by patient referral and during clinical checks.

CONTACTS AND LOCATIONS:
Overall Officials: Felice Roberto Grassi, PhD, Principal Investigator — University of Bari
Locations (1):
- Aldo Moro University, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared with researchers who make an official request

REFERENCES:
- [Background] Lima de Andrade C, Carvalho MA, Bordin D, da Silva WJ, Del Bel Cury AA, Sotto-Maior BS. Biomechanical Behavior of the Dental Implant Macrodesign. Int J Oral Maxillofac Implants. 2017 Mar/Apr;32(2):264-270. doi: 10.11607/jomi.4797. PMID 28291847
- [Background] Cali M, Zanetti EM, Oliveri SM, Asero R, Ciaramella S, Martorelli M, Bignardi C. Influence of thread shape and inclination on the biomechanical behaviour of plateau implant systems. Dent Mater. 2018 Mar;34(3):460-469. doi: 10.1016/j.dental.2018.01.012. Epub 2018 Feb 1. PMID 29395470
- [Background] Grassi FR, Grassi R, Rapone B, Alemanno G, Balena A, Kalemaj Z. Dimensional changes of buccal bone plate in immediate implants inserted through open flap, open flap and bone grafting and flapless techniques: A cone-beam computed tomography randomized controlled clinical trial. Clin Oral Implants Res. 2019 Dec;30(12):1155-1164. doi: 10.1111/clr.13528. Epub 2019 Sep 11. PMID 31461183
- [Result] Scarano A, Assenza B, Inchingolo F, Mastrangelo F, Lorusso F. New Implant Design with Midcrestal and Apical Wing Thread for Increased Implant Stability in Single Postextraction Maxillary Implant. Case Rep Dent. 2019 Sep 5;2019:9529248. doi: 10.1155/2019/9529248. eCollection 2019. PMID 31583139